CLINICAL TRIAL: NCT06442319
Title: The Efficiency and Safety of Platelet-rich Plasma Intra-articular Injections After Anterior Cruciate Ligament Reconstruction: MRI and Clinical Outcome Analysis.
Brief Title: The Efficiency and Safety of PRP Treatment After Anterior Cruciate Ligament Reconstruction.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nicolaus Copernicus University in Toruń, Collegium Medicum in Bydgoszcz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NicolausCopernicusU
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: ACL Injury; Knee Osteoarthritis; Knee Injuries
Keywords: PRP, ACL reconstruction, knee osteoarthritis
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Osteoarthritis, Knee; Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet-rich Plasma (Experimental)
  Interventions: Biological: Platelet-rich plasma
- Hyaluronic Acid (Active Comparator)
  Interventions: Biological: Platelet-rich plasma

INTERVENTIONS:
Biological: Platelet-rich plasma — Platelet-rich plasma intra-articular injection in patients after anterior cruciate ligament reconstruction

SUMMARY:
The anterior cruciate ligament (ACL) is the main stabilizer of the knee joint, as it controls anteroposterior and rotatory knee laxity. The number of ACL injuries has increased in the past three decades because more and more people participate in recreational and competitive sporting activities. Injury to the ACL often leads to functional instability, damage to the meniscus and articular cartilage, and an increased risk for osteoarthritis (OA). Emphasizes the fact that ACL has limited healing potential 'The gold standard' treatment is ACL reconstruction, with over 200,000 reconstruction surgeries performed annually in the United States. However, despite the success of surgery in restoring functional stability, it has been found so far in several studies that the prevalence of moderate to severe arthritis in long-term radiographic follow-up is more than 50% after ACL reconstruction within 5 to 15 years or sooner. ACL-injured knees had at least 3 times higher risk of arthritis than uninjured contralateral knees. Early osteoarthritis was observed on magnetic resonance imaging (MRI) up to 11 years following ACL injury after operative and nonoperative management. Because ACL injuries predominantly occur in individuals between the ages of 15 and 25 years, symptoms of OA most often affect patients during their most productive years. This is worrisome because most patients who sustain ACL tears are free of the risk of other factors for developing OA.Consequently, posttraumatic OA after ACL reconstruction ultimately translates into a large economic effect on the healthcare system owing to the young age of this population. Platelet-rich plasma is an autologous solution of highly concentrated platelets dispersed in a small capacity of plasma. Enthusiasm for the therapeutic potential of platelets is based on its rich omplement of anabolic growth factors and anti-inflammatory cytokines in the platelets, which induce cellular proliferation, migration, differentiation, angiogenesis, and extracellular matrix synthesis. In addition, the functional mechanisms of PRP in OA treatment have been explained by its effect on modulating critical pro-inflammatory mediators and catabolic enzymes, as well as maintaining joint homeostasis. The reasons for this early incidence of post-traumatic OA remain unclear, but the underlying mechanisms have been speculated to involve some combination of cartilage damage at the time of injury, and posttraumatic molecular changes in the joint, including immune reactions or persistent secondary inflammation. We hypothesized that PRP injection after ACL reconstruction could prevent cartilage damage, act anti-inflammatory, and provide better clinical and radiological outcomes seen in MRI.

ELIGIBILITY:
Inclusion Criteria:

* subject is 18-45 years old
* subject has BMI < 40 kg/m2
* subject had ACL reconstrution
* small asymptomatic meniscal lesions that won't require repair
* subject must be willing to abstain from other intra-articular treatments of the knee for the duration of the study.
* subject is willing to discontinue all analgesics including nonsteroidal anti-inflammatory drugs (NSAIDs), except tramadol and paracetamol, at least one month before the synovial fluid aspiration and through the completion of the study
* subject is able to understand and comply with the requirements of the study and voluntarily provides consent

Exclusion Criteria:

* subject has a history of metabolic diseases, endocrine disorders, rheumatic and connective tissue diseases, cancer, hormonal contraception, steroid therapy, antibiotic therapy
* subject had an intraarticular injection into the affected joint
* subject had previous operations (beside ACL reconstruction) or fractures of the affected limb
* subject has a history of nicotine, alcohol, or drug addiction
* subject has a meniscal tear that requires suturing or total meniscectomy seen on MRI
* subject has multi-ligament knee injuries or multi-organ injury
* subject has significant varus or valgus deformity greater than 10 degrees in either knee, determined by an X-ray

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2028-04-15 (Estimated); Study Completion 2030-04-15 (Estimated)

PRIMARY OUTCOMES:
Pain and cartilage volume | 12 months
  The 2 primary outcomes were 12-month change in overall average knee pain scores (11-point scale; range, 0-10, with higher scores indicating worse pain; minimum clinically important difference of 1.8) and percentage change in cartilage volume as assessed by magnetic resonance imaging (MRI).

SECONDARY OUTCOMES:
Synovitis | 6 and 12 months post-treatment
  The assesment of synovial fluid volume and fat pad synovitis seen in ultrasonography and MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Dawid Szwedowski, Torun, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lohmander LS, Ostenberg A, Englund M, Roos H. High prevalence of knee osteoarthritis, pain, and functional limitations in female soccer players twelve years after anterior cruciate ligament injury. Arthritis Rheum. 2004 Oct;50(10):3145-52. doi: 10.1002/art.20589. PMID 15476248
- [Background] Frobell RB, Roos EM, Roos HP, Ranstam J, Lohmander LS. A randomized trial of treatment for acute anterior cruciate ligament tears. N Engl J Med. 2010 Jul 22;363(4):331-42. doi: 10.1056/NEJMoa0907797. PMID 20660401